CLINICAL TRIAL: NCT04803513
Title: Observational Study on the Efficacy, Safety, and Tolerability of GAlcanezumab in Real Life Migraine Patients in ITaly (GARLIT)
Brief Title: Observational Study on the Efficacy, Safety, and Tolerability of GAlcanezumab in Real Life Migraine Patients in ITaly
Acronym: GARLIT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Sponsor
Other Study IDs: GARLIT; IRB Number (Registry Identifier: 30/20 OSS)
Record Dates: First submitted 2021-03-09; First posted 2021-03-17 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — galcanezumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Galcanezumab — Galcanezumab according to clinical indication in real life

SUMMARY:
Objective: To determine in real life the efficacy, safety and tolerability of galcanezumab in the prevention of high-frequency episodic migraine (HFEM) and chronic (CM) migraine.

Design: This prospective observational cohort study was conducted between November 2019 and January 2021.

Participants: Consecutive adult HFEM and CM patients clinically prescribed galcanezumab were enrolled.

Setting: Multicenter study in 13 Italian headache centers.

Exposure: Galcanezumab subcutaneous injection 120 mg monthly with the first loading dose of 240 mg.

Main Outcome(s) and Measure(s): The primary end-point was the change in monthly migraine days (MMDs) in HFEM patients and monthly headache days (MHDs) in CM ones after six months of therapy (V6) compared to baseline. Secondary end-points included variation in Numerical Rating Scale (NRS), monthly painkiller intake (MPI), HIT-6, and MIDAS scores. We assessed 50%, 75%, and 100% responder rates (RR), the conversion rate from CM to episodic migraine (EM), and the Medication Overuse condition to the non-overuser.

DETAILED DESCRIPTION:
GARLIT is an independent, multicenter, prospective, cohort, real-life study. All consecutive patients aged 18 or older with a diagnosis of HFEM (8-14 migraine days per month) or CM (1.3 ICHD-3), who had failed at least three migraine preventive treatments and not previously involved in any CGRP mAbs trial, are considered for enrolment. Patients are assessed at baseline by a headache expert neurologist with a face-to-face interview using a semi-structured questionnaire addressing socio-demographic factors, clinical migraine features, previous and current acute and preventive migraine treatments, comorbidities and concomitant medications. Headache-related dopaminergic and autonomic symptoms, temporal artery turgidity/hyperpulsatility, and allodynia during or between attacks are also investigated. Patients are also requested to rate the overall efficacy of triptans in most attacks as none/poor (0) or fair/excellent (1).

Enrolled patients will carefully fill in a headache diary during a run-in month period (baseline) and the entire duration of the study, to report monthly migraine days (MMDs) for HFEM patients, all monthly headache days (MHDs) of at least moderate intensity for CM subjects, and monthly painkillers intake (MPI). Patients were also asked to rate pain severity (using the 0-10 Numerical Rating Scale, NRS) of the worst painful attack and fill in migraine disability questionnaires (Headache Impact Test, HIT-623, monthly, and the MIgraine Disability Assessing Scale24, MIDAS, quarterly).

Patients will be treated with galcanezumab subcutaneous injection with the first loading dose of 240mg and then every month with 120mg as recommended, according to real life clinical indication (www.europa.ema.eu).

The above-reported variables and any adverse event (AE) are recorded at baseline and monthly at every in-office visits. Telephone/email contacts are allowed when in-office visits are not possible. All AEs are reported to Eudravigilance and classified as gastrointestinal (e.g. nausea, constipation), cutaneous (e.g. injection-site reactions: rash/erythema, pruritus, urticaria, oedema/induration), arthralgia, Raynaud phenomenon, dizziness and other (<1% of patients: i.e. somnolence, alopecia, anxiety).

Patients will provide written informed consent.

ELIGIBILITY:
Inclusion Criteria:

* the clinical indication for Galcanezumab as a preventive treatment for Migraine according to European Medicines Agency
* age18 years or older
* 8 or more mean Monthly Migraine Headache days in the last three months

Exclusion Criteria:

- previous exposure to any monoclonal antibodies inhibiting CGRP pathway, including clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients aged 18 or older with a diagnosis of high-frequency episodic migraine (8-14 migraine days per month) or chronic migraine (1.3 ICHD-3),
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
e change in monthly migraine days (MMDs) on galcanezumab therapy compared to baseline | baseline, monthly and through therapy cycle completion which is an average of 1 year. and after three months after therapy withdrawal.
  MMDs defined as monthly migraine days collected by headache diary

SECONDARY OUTCOMES:
variation in Numerical Rating Scale (NRS), monthly painkiller intake (MPI) during galcanezumab therapy compared to baseline | baseline, monthly and through therapy cycle completion, which is an average of 1 year, and after three months after therapy withdrawal.
  NRS= 0-to-10 pain intensity of the worst migraine attacks perceived in the previous month, MPI= the number of painkiller taken in the previous month.

CONTACTS AND LOCATIONS:
Overall Officials: Fabrizio Vernieri, MD, Principal Investigator — Campus Bio-Medico University
Locations (1):
- Campus Bio Medico University Hospital, Rome, RM, Italy

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be shared upon request to any qualified investigator

REFERENCES:
- [Derived] Altamura C, Brunelli N, Marcosano M, Aurilia C, Egeo G, Lovati C, Favoni V, Perrotta A, Maestrini I, Schiano Di Cola F, d'Onofrio F, Finocchi C, Bertuzzo D, Bono F, Ranieri A, Albanese M, Messina R, Doretti A, Di Piero V, Cevoli S, Barbanti P, Vernieri F; GARLIT Study Group. Conversion from chronic to episodic migraine in patients treated with galcanezumab in real life in Italy: the 12-month observational, longitudinal, cohort multicenter GARLIT experience. J Neurol. 2022 Nov;269(11):5848-5857. doi: 10.1007/s00415-022-11226-4. Epub 2022 Jun 28. PMID 35763113
- [Derived] Vernieri F, Altamura C, Brunelli N, Costa CM, Aurilia C, Egeo G, Fofi L, Favoni V, Lovati C, Bertuzzo D, d'Onofrio F, Doretti A, Di Fiore P, Finocchi C, Schiano Di Cola F, Ranieri A, Colombo B, Bono F, Albanese M, Cevoli S, Barbanti P; GARLIT Study Group. Rapid response to galcanezumab and predictive factors in chronic migraine patients: A 3-month observational, longitudinal, cohort, multicenter, Italian real-life study. Eur J Neurol. 2022 Apr;29(4):1198-1208. doi: 10.1111/ene.15197. Epub 2021 Dec 6. PMID 34826192
- [Derived] Vernieri F, Altamura C, Brunelli N, Costa CM, Aurilia C, Egeo G, Fofi L, Favoni V, Pierangeli G, Lovati C, Aguggia M, d'Onofrio F, Doretti A, Di Fiore P, Finocchi C, Rao R, Bono F, Ranieri A, Albanese M, Cevoli S, Barbanti P; GARLIT Study Group. Galcanezumab for the prevention of high frequency episodic and chronic migraine in real life in Italy: a multicenter prospective cohort study (the GARLIT study). J Headache Pain. 2021 May 3;22(1):35. doi: 10.1186/s10194-021-01247-1. PMID 33941080